CLINICAL TRIAL: NCT00619112
Title: Phase II Study of 7 Days On/7 Days Off Temozolomide in Patients With High-Grade Glioma
Brief Title: Temozolomide in Treating Patients With Recurrent High-Grade Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSF-07107; SPRI-UCSF-H44867-31182-01; NCT00539552 (obsolete NCT alias)
Record Dates: First submitted 2008-02-19; First posted 2008-02-20 (Estimated); Results first posted 2013-10-29 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Recurrent Central Nervous System Neoplasm
Keywords: adult glioblastoma; adult gliosarcoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult mixed glioma; recurrent adult brain tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma; Astrocytoma; Oligodendroglioma; Glioma; Brain Neoplasms | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Temozolomide (Experimental): single arm trial; Patients treated with temozolomide at a dose of 150mg/m2 daily for seven consecutive days of every other week. One 28-day cycle will include treatment with temozolomide on days 1-7 and days 15-21 with no treatment on days 8-14
  Interventions: Drug: temozolomide

INTERVENTIONS:
Drug: temozolomide — single arm study
  Other Names: temodar

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well temozolomide works in treating patients with recurrent high-grade glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy, as measured by 6-month progression-free survival, of a dose-intense temozolomide treatment schedule in patients with recurrent high-grade glioma.

Secondary

* Assess the toxicities of this dose-intense temozolomide.
* Determine the overall survival of patients treated with this dose-intense schedule.
* Determine whether methylation status of the MGMT gene within patients' tumors predicts greater efficacy (progression-free survival), in patients treated on this protocol.
* Determine whether patients' tumors have functional alterations of the mismatch repair (MMR) system by PCR analysis for microsatellite instability (MSI) and whether such alterations may influence outcome in patients treated on this protocol.
* Determine how initial success with temozolomide may influence outcome in recurrent patients treated on this protocol by evaluating patients progressing after two first-line adjuvant courses of temozolomide, patients progressing within 6 months after the 6th adjuvant course of temozolomide, and patients progressing 6 months after temozolomide is voluntarily discontinued.

OUTLINE: Patients receive oral temozolomide once daily on days 1-7 and days 15-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Formalin-fixed paraffin-embedded tissue blocks or unstained paraffin slides from available surgical samples are evaluated for molecular abnormalities in the tumor, including (but not limited to) MGMT status and microsatellite instability.

After completion of study therapy, patients are followed every 3 months for survival.

PROJECTED ACCRUAL: A total of 40 patients with WHO II grade 4 tumors (glioblastoma multiforme [GBM]) and 20 patients with WHO II grade 3 tumors (non-GBM) will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria

* Patients with radiographically proven recurrent, intracranial malignant glioma will be eligible for this protocol.
* All patients must sign an informed consent
* Patients must have had external beam radiation; there is no limit to the number of prior chemotherapies used.
* Patients must be > 18 years old, and with a life expectancy > 8 weeks.
* Patients must have a Karnofsky performance status of > 60.
* At the time of registration: Patients must have recovered from the toxic effects of prior therapy:
* Patients must have adequate bone marrow function.
* Patients must have shown unequivocal radiographic evidence for tumor progression by MRI
* Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as all of the following conditions apply: They have recovered from the effects of surgery. Residual disease following resection of recurrent intracranial malignant glioma is not mandated for eligibility into the study.
* Patients must have failed prior radiation therapy and must have an interval of greater than or equal to 42 days from the completion of radiation therapy to study entry.
* Patients with prior therapy that included interstitial brachytherapy, stereotactic radiosurgery, or Gliadel wafers must have confirmation of true progressive disease rather than radiation necrosis based upon either PET or MR spectroscopy or surgical documentation of disease.
* Male and female patients with reproductive potential must use an approved contraceptive method

Exclusion Criteria

* Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy
* Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible.
* Patients must not have active infection or serious intercurrent medical illness.
* Patients must not be pregnant/breast feeding and must agree to practice adequate contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-10; Primary Completion 2011-12 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas A. Butowski, MD, Principal Investigator — University of California, San Francisco; Susan M. Chang, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States

REFERENCES:
- [Derived] Han SJ, Rolston JD, Molinaro AM, Clarke JL, Prados MD, Chang SM, Berger MS, DeSilva A, Butowski NA. Phase II trial of 7 days on/7 days off temozolmide for recurrent high-grade glioma. Neuro Oncol. 2014 Sep;16(9):1255-62. doi: 10.1093/neuonc/nou044. Epub 2014 Mar 26. PMID 24670608

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from within established neuro oncology clinic at UCSF. First paient 11.5.2007 and last patient 1.24.2012
Groups:
- Glioblastoma: Glioblastoma patients were treated with temozolomide at a dose of 150mg/m^2 daily for seven consecutive days of every other week.
  One 28-day cycle included treatment with temozolomide on days 1-7 and days 15-21 with no treatment on days 8-14
- Grade III Glioma: Grade III glioma patients were treated with temozolomide at a dose of 150mg/m^2 daily for seven consecutive days of every other week.
  One 28-day cycle included treatment with temozolomide on days 1-7 and days 15-21 with no treatment on days 8-14
Period: Overall Study
Arm/Group | Glioblastoma | Grade III Glioma
Started | 40 | 20
Completed | 39 (Data from patient who didn't complete study was still included in the final analysis.) | 18 (Data from patients who didn't complete study was still included in the final analysis.)
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glioblastoma | Grade III Glioma | Total
Number analyzed (Participants) | 40 | 20 | 60
Age, Continuous [Median (Full Range); unit: years] | 55 [30 to 68] | 48 [27 to 70] | 53 [27 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 28 | 10 | 38
Region of Enrollment [Number; unit: participants]
  United States | 40 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: 6 Month Progression-free Survival
Description: Efficacy of dose-intense temozolomide treatment schedule, as measured by 6 months progression-free survival
Time Frame: First day of treatment until progression or until 6 months mark
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Glioblastoma | Grade III Glioma
Number analyzed (Participants) | 40 | 20
percentage of patients | 10 [3 to 24] | 50 [27 to 73]

2. Secondary Outcome: Progression-free Survival (PFS) Based on Tumor MGMT (O(6)-Methylguanine-DNA Methyltransferase) Promoter Methylation Status.
Description: Progression-free survival data (obtained for Primary Outcome Measure) was correlated with tumor MGMT (O(6)-methylguanine-DNA methyltransferase) promoter methylation status, obtained from patients as part of the study.
Time Frame: First day of treatment until progression or until 6 months mark
Population: Tumor tissue was available for the exploratory MGMT methylation analysis in 48 patients. In 7 samples the tissue was inadequate for analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Glioblastoma With Methylated MGMT: PFS of Glioblastoma patients with methylated MGMT tumors
- Glioblastoma With Unmethylated MGMT: PFS of Glioblastoma patients with unmethylated MGMT tumors
- Grade III Glioma With Methylated MGMT: PFS of Grade III Glioma patients with methylated MGMT tumors
- Grade III Glioma With Unmethylated MGMT: PFS of Grade III Glioma patients with unmethylated MGMT tumors
Arm/Group | Glioblastoma With Methylated MGMT | Glioblastoma With Unmethylated MGMT | Grade III Glioma With Methylated MGMT | Grade III Glioma With Unmethylated MGMT
Number analyzed (Participants) | 7 | 21 | 10 | 3
weeks | 8.14 [7.71 to NA] — Upper confidence limit for median cannot be estimated (not yet reached). | 7.57 [7.29 to 9] | 38.1 [10.71 to NA] — Upper confidence limit for median cannot be estimated (not yet reached). | 48.6 [6.86 to NA] — Upper confidence limit for median cannot be estimated (not yet reached).

3. Secondary Outcome: Overall Survival
Time Frame: up to 2 years after treatment
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Glioblastoma | Grade III Glioma
Number analyzed (Participants) | 40 | 20
weeks | 21.6 [16.9 to 30.6] | 100.6 [67 to NA] — The upper bound was not reached during length of the study.

4. Secondary Outcome: Patients With Tumors With Functional Alterations of the Mismatch Repair (MMR) System
Description: PCR analysis of tumor tissue for microsatellite instability (MSI). Tissue was obtained during surgeries prior this study.
Time Frame: prior to start of study
Measure: Count of Participants; unit: Participants
Arm/Group | Glioblastoma | Grade III Glioma
Number analyzed (Participants) | 40 | 20
Participants | 0 | 0

5. Secondary Outcome: Patients Progressing After Two First-line Adjuvant Courses of Temozolomide
Time Frame: After two first-line adjuvant courses of temozolomide
Measure: Count of Participants; unit: Participants
Arm/Group | Glioblastoma | Grade III Glioma
Number analyzed (Participants) | 40 | 20
Participants | 3 | 0

6. Secondary Outcome: Patients Progressing Within 6 Months After 6th Adjuvant Course of Temozolomide
Time Frame: Within 6 months after 6th adjuvant course of temozolomide
Measure: Count of Participants; unit: Participants
Arm/Group | Glioblastoma | Grade III Glioma
Number analyzed (Participants) | 40 | 20
Participants | 4 | 1

7. Secondary Outcome: Patients Progressing 6 Months After Temozolomide is Voluntarily Discontinued
Time Frame: From beginning of voluntarily temozolomide discontinued up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Glioblastoma | Grade III Glioma
Number analyzed (Participants) | 40 | 20
Participants | 4 | 4

ADVERSE EVENTS:
Arm/Group | Temozolomide
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 38/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Temozolomide (N=60)
Lymphocyte count decreased (Investigations) | 28
White blood cell decreased (Investigations) | 7
Neutrophil count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 4
Peripheral motor neuropathy (Nervous system disorders) | 6
Depressed level of consciousness (Nervous system disorders) | 3
Seizure (Nervous system disorders) | 2
Dysphasia (Nervous system disorders) | 2
Confusion (Psychiatric disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Fatigue (General disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pain (General disorders) | 2
Skin infection (Infections and infestations) | 1
Eye disorders - Other, specify (Eye disorders) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1

LIMITATIONS AND CAVEATS:
The trial reached enrollment. There were no unexpected toxicities.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No